CLINICAL TRIAL: NCT05105412
Title: A Single Arm，Phase Ib/II Study of the Combination of Lenalidomide and Gemcitabine in Relapsed or Refractory Peripheral T-cell Lymphomas (PTCL)
Brief Title: Lenalidomide and Gemcitabine in Relapsed or Refractory Peripheral T-cell Lymphomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The resolution of DSMB
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); National Cheng-Kung University Hospital (Other); China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1421
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Peripheral T-cell Lymphomas (PTCL)
Keywords: peripheral T-cell lymphomas (PTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Lenalidomide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide and Gemcitabine (Experimental): Lenalidomide and Gemcitabine
  Interventions: Drug: Lenalidomide and Gemcitabine (Dose level 11); Drug: Lenalidomide and Gemcitabine (Dose level 21); Drug: Lenalidomide and Gemcitabine (Dose level 31); Drug: Lenalidomide and Gemcitabine (Dose level 41)

INTERVENTIONS:
Drug: Lenalidomide and Gemcitabine (Dose level 11) — lenalidomide 25 mg/day D1-D14 and gemcitabine 1000 mg/m2 D1, D8
  Other Names: Dose level 11
Drug: Lenalidomide and Gemcitabine (Dose level 21) — lenalidomide 15 mg/day D1-D14 and gemcitabine 1000 mg/m2 D1, D8
  Other Names: Dose level 21
Drug: Lenalidomide and Gemcitabine (Dose level 31) — lenalidomide 10 mg/day D1-D14 and gemcitabine 1000 mg/m2 D1, D8
  Other Names: Dose level 31
Drug: Lenalidomide and Gemcitabine (Dose level 41) — lenalidomide 10 mg/day D1-D14 and gemcitabine 800 mg/m2 D1, D8
  Other Names: Dose level 41

SUMMARY:
This is a single country multi-center, open-label phase Ib/II single-arm study in relapsed or refractory PTCL patients. Patients will be treated with the combination of lenalidomide and gemcitabine until disease progression, intolerable toxicity, or patient withdrawal.

DETAILED DESCRIPTION:
There are 3000 newly diagnosed lymphoma patients in Taiwan, and T-cell neoplasms accounted for 17.4% of total lymphomas. Peripheral T-cell lymphomas (PTCL) are heterogeneous malignancies, and peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), and anaplastic large cell lymphoma (ALCL) are the most common subtypes.

Patients with relapsed or refractory PTCL to 1st-line chemotherapy had dismal prognosis under conventional chemotherapy. Combination of gemcitabine with platinum chemotherapy may be effective regimens, because they provided objective response rate (ORR) of 70% in PTCL patients. Since most salvage chemotherapy regimens provided limited activity in PTCL, many new regimens were studied in PTCL. Except brentuximab vedotin provided high activity through targeting CD30 on ALCL, new regimens (including lenalidomide) provided ORR about 20% and PFS about 3 months in PTCL.

Lenalidomide is an immunomodulatory agent, and it reduces T-regulatory cells, activates CD8-positive T cells, and increases natural killer cell numbers and in activation status. Gemcitabine may augment immune responses in several ways: activating T cells, increasing the amount of dendritic cells, increasing the amounts of antigens loaded onto antigen-presenting cells, and down-regulating T-regulatory cells. We design this phase 2 study under the hypothesis of synergistic effect of anti-tumor immunity and efficacy to PTCL in combination with lenalidomide and gemcitabine. The dose of lenalidomide monotherapy to treat PTCL is 25 mg daily based on previous studies, and we also start this dose in our study initially. Lenalidomide in combination with gemcitabine in 1st-line treatment of patients with advanced pancreatic cancer were studied before. Patients could tolerate oral lenalidomide of 25 mg daily on days 1 to 21, and intravenous gemcitabine dose of 1000 mg/m2 on days 1, 8, and 15, of each 28-day cycle. Because our enrolled patients will receive previous-line chemotherapy and combination of lenalidomide and gemcitabine may exacerbate myelosuppression, we designed oral lenalidomide of 25 mg daily on days 1 to 14, and intravenous gemcitabine dose of 1000 mg/m2 on days 1 and 8, of each 21-day cycle. In order to monitor toxicities and adjust drug doses closely, we arrange phase Ib study to evaluate dose-limiting toxicities about combination of lenalidomide and gemcitabine. The schedules about dose delays and modifications were also designed in phase Ib and II studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (20 years of age) have the following three subtypes of PTCL:

(1)Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS), (2)Angioimmunoblastic lymphoma (AITL), or (3)Anaplastic large cell lymphoma (ALCL). If patients had CD30-positive systemic ALCL, they should receive brentuximab vedotin before enrollment 2. (1) In transplant-eligible patients: patients who have relapsed disease after autologous stem-cell transplantation (2) In transplant-ineligible patients: patients who have received at least first-line systemic chemotherapy treatment and have a stable disease, progressive disease, or relapsed disease.

3. Patients have an ECOG Scale of Performance Status score of 0-1. 4. Patients have at least one measurable lesion by CT with a size of > 1.5 cm in at least one axis.

5. Patients have adequate renal function: serum creatinine (Cr) ≤ 1.5 times the upper limit of normal range (ULN) and calculated creatinine clearance (Ccr) ≥ 40 mL/min.

6. Patients have adequate bone marrow function:

1. Absolute neutrophil count (ANC) ≥ 1500/μL, Without growth factor support (filgrastim or lenograstim) for at least 14 days
2. Platelet count ≥ 75 000/μL. Evaluated at least 7 days after last platelet transfusion
3. Hemoglobin ≥ 8 g/dL. May receive transfusion 7. Patients have adequate hepatic function: serum alkaline phosphatase (ALP), alanine, or aspartate aminotransferase levels (ALT & AST) ≤ 2.5 times the ULN and serum total bilirubin ≤ 1.5 times the ULN.

Exclusion Criteria:

1. Patients have already been exposed to lenalidomide and gemcitabine.
2. Patients have less than 100 days from previous autologous stem cells transplantation prior to first study drug dose.
3. Patients have HIV infection.
4. Patients have cerebral or meningeal disease including signs or symptoms of progressive multifocal leukoencephalopathy.
5. Patients have symptomatic neurologic disease compromising normal activities of daily living or requiring medication.
6. Patients have any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose.
7. Patients received prior immunosuppressive chemotherapy, therapeutic radiation, or any immunotherapy (eg, immunoglobulin replacement, other monoclonal antibody therapies) within 4 weeks of first study drug dose.
8. Patients have known hypersensitivity to any excipient contained in the drug formulation of lenalidomide or gemcitabine.
9. Patients have known positive hepatitis B surface antigen but not receive anti-hepatitis B drug, or known or suspected active hepatitis B and C infection.
10. Patients have diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
11. Patients have any of the following cardiovascular conditions or values within 6 months before the first dose of study drug:

    * A left-ventricular ejection fraction <50%.
    * Myocardial infarction within 2 years of randomization.
    * New York Heart Association (NYHA) Class III or IV heart failure
    * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
12. Patients with unstable medical or psychiatric conditions or a history of any other serious medical disease deemed inappropriate for inclusion in this study, as determined by the investigators.
13. Women who are pregnant or breastfeeding or have a positive pregnancy test during screening or Day 1 before the first dose of study drug.
14. Women of childbearing potential who do not use two effective contraceptive methods from the time of signing informed consent through 6 months after the last dose of study drug or agree to completely abstain from heterosexual intercourse.
15. Male patients, even if surgically sterilized, (i.e., status post vasectomy) who do not agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
16. Patients with a life expectancy of <3 months, as determined by the investigators.
17. Patients with, as judged by the investigators, other contraindications for lenalidomide and gemcitabine administration, such as concurrent usage of drugs that may have potentially severe drug-drug interactions.
18. Patients who are unwilling or unable to give consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
DLT | 12 months
  To evaluate the dose-limited toxicity (DLT) of combination of lenalidomide and gemcitabine
ORR | 24 months
  To evaluate the objective response rate of combination of lenalidomide and gemcitabine by Lugano classification

SECONDARY OUTCOMES:
PFS | 24months
  To evaluate the progression free survival of combination of lenalidomide and gemcitabine by Lugano classification
OS | 24months
  To evaluate the overall survival of combination of lenalidomide and gemcitabine by Lugano classification
Treatment-related adverse events | 24months
  To evaluate the number of participants with treatment-related adverse events assessed by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, Study Director — Taiwan Cooperative Oncology Group, NHRI
Locations (5):
- Taiwan (5):
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei